CLINICAL TRIAL: NCT03815682
Title: A Phase 1/2 Study of Deep IL-15 Loaded T-Cells Alone and in Combination With Pembrolizumab in Patients With Select Solid Tumors and Lymphomas
Brief Title: RPTR-147 in Patients With Selected Solid Tumors and Lymphomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Development program terminated
Sponsor: Repertoire Immune Medicines (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TT-101; KEYNOTE KN-948 (Other: Merck)
Record Dates: First submitted 2019-01-14; First posted 2019-01-24 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Solid Tumor; Lymphoma
Keywords: HPV-16 E6/E7 positive solid tumors; Melanoma
MeSH Terms: conditions — Lymphoma; Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- RPTR-147:1 (Experimental): Arm A: Escalating doses of RPTR-147:1 as a monotherapy in solid tumors and lymphomas
  Interventions: Biological: Arm A: RPTR-147:1
- RPTR-147:1 and Pembrolizumab (Experimental): Arm B: Escalating doses of RPTR-147:1 in combination with Pembrolizumab in patients with solid tumors and lymphomas
  Interventions: Biological: Arm B: RPTR-147:1 and Pembrolizumab
- RPTR-147:2 (Experimental): Arm C: Escalating doses of RPTR-147:2 in patients with HPV-16 positive tumors
  Interventions: Biological: Arm C: RPTR-147:2

INTERVENTIONS:
Biological: Arm A: RPTR-147:1 — Escalating doses of RPTR-147:1 as a monotherapy
  Arms: RPTR-147:1
Biological: Arm B: RPTR-147:1 and Pembrolizumab — Escalating doses of RPTR-147:1 in combination with Pembrolizumab
  Arms: RPTR-147:1 and Pembrolizumab
Biological: Arm C: RPTR-147:2 — Escalating doses of RPTR-147:2 in patients with HPV positive tumors
  Arms: RPTR-147:2

SUMMARY:
The purpose of this study is to assess the safety and tolerability of escalating doses of RPTR-147 as a monotherapy and in combination with Pembrolizumab in patients with selected solid tumors and lymphomas.

DETAILED DESCRIPTION:
This is a first-in-human, open-label, multicenter, dose escalation study designed to determine the safety and tolerability of RPTR-147 as a monotherapy and in combination with Pembrolizumab in patients with selected solid tumors or lymphomas.

The study will include 2 dosing periods: A Dose Escalation (Phase 1) followed by an Expansion (Phase 2).

ELIGIBILITY:
INCLUSION CRITERIA:

Patients eligible for inclusion in this study must meet all of the following criteria:

1. Be willing and able to provide written informed consent for the trial.
2. Written informed consent must be obtained prior to any study procedures.
3. Age ≥18 years (or ≥16 years at Dana Farber Cancer Institute).
4. Histologically- or cytologically-confirmed relapsed/refractory metastatic or locally-advanced solid tumor or lymphoma whose disease has progressed despite all appropriate curative or life-prolonging treatments, are intolerant to these therapies or have refused standard treatment.

   1. Inclusion criteria: RPTR-147:1 (Arms A & B) treatment groups

      Cohort enrollment may be limited to potentially immune-responsive tumor types meeting the above criterion during the first approximately 2 weeks of the enrollment period of each cohort due to their potential to respond to and activate RPTR-147:1:
      * NSCLC
      * Melanoma
      * Clear cell cancer of the kidney
      * HNSCC
      * Urothelial cancer
      * Lymphoma
      * Sarcomas
      * Ovarian Cancer
      * Based upon emerging data that will be discussed during the Safety Review Committee meetings, the patient population may be further limited based other factors
   2. Inclusion criteria: RPTR-147:2 (Arm C) treatment group Patients with cancers known to be HPV-16 positive.
5. Patient must have documented HLA-typing results that meet the study requirements. The list of eligible HLA alleles will be updated on an ongoing basis by the Sponsor.

   • Once sufficient data has been collected for drug product analytics, or sufficient HLA coverage is obtained, the HLA-type eligibility requirement may be discontinued by the Sponsor.
6. For patients with solid tumors, use Response Evaluation Criteria in Solid Tumor (RECIST) v1.1: measurable disease (at least one measurable non-nodal lesion of at least 1.0 cm in longest diameter or nodal lesion of at least 1.5 cm in shortest diameter) documented within 10 weeks of their projected C1D1 visit.

   For patients with lymphoma, use the Lugano classification: measurable disease defined as at least one lesion that can be accurately measured in at least two dimensions with spiral computed tomography (CT) scan documented within 10 weeks of their projected C1D1 visit. Minimum measurement must be >15 mm in the longest diameter.

   NOTE: If there are no pre-existing radiologic assessments within 10 weeks of the projected C1D1 visit, other evidence of measurable disease may be considered sufficient to fulfill this criterion following documented discussion and approval from the Sponsor.

   NOTE: Please note, for dosing/Screening Period 2, patients must have a radiological assessment per mRECIST v1.1 (solid tumor) or Lugano classification (lymphomas) within 28 days before receiving treatment with RPTR-147 to serve as the patient's baseline tumor assessment.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1.
8. Have provided archival tumor tissue sample or newly obtained core or excisional biopsy, during screening period 2, of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue. Further details can be found in the Laboratory Manual.

   Note: If submitting unstained cut slides, newly cut slides should be submitted to the testing laboratory within 14 days from the date slides are cut.
9. RPTR-147:1 in combination with pembrolizumab (Arm B only) - Patients should have malignancies for which the response rate to anti-PD1/PDL1 monotherapy is <20% or, if they have malignancies for which anti-PD1/PDL1 are standard of care must have progressed on treatment with an anti-PD1/L1 monoclonal antibody (mAb) administered either as monotherapy, or in combination with other checkpoint inhibitors or other therapies. PD-1 treatment progression is defined by meeting all of the following criteria:

   1. Has received at least 2 doses of an approved anti-PD-1/L1 mAb.
   2. Has demonstrated disease progression (PD) after PD-1/L1 as defined by RECIST v1.1. The initial evidence of PD is to be confirmed by a second assessment no less than four weeks from the date of the first documented PD, in the absence of rapid clinical progression.
   3. Progressive disease has been documented as per the following within 12 weeks from the last dose of anti-PD-1/L1 mAb.
10. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    1. Not a woman of childbearing potential (WOCBP)
    2. A WOCBP who agrees to follow contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment.
11. A male participant must agree to use contraception during the treatment period and for at least 165 days after the last dose of study treatment.

EXCLUSION CRITERIA:

Patients eligible for this study must not meet any of the following criteria:

1. Previously identified hypersensitivity to components of RPTR-147 or excipients.
2. Pembrolizumab combination Arm B only - Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
3. Patients with T-cell lymphomas or small lymphocytic lymphoma.
4. Presence of active central nervous system (CNS) disease and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable, and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
5. Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease. For any interim radiotherapy received after the baseline tumor assessment, the target lesions must not be irradiated.
6. Patient having out of range laboratory values defined as:

   * Creatinine clearance (calculated using Cockcroft-Gault formula, or measured) <40 mL/min
   * Total bilirubin >1.5 x upper limit of normal (ULN), except for patients with Gilbert's syndrome who are excluded if total bilirubin >3.0 x ULN or direct bilirubin >1.5 x ULN
   * Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) >3 x ULN, except for patients that have tumor involvement of the liver, who are excluded if ALT >5 x ULN
   * Absolute neutrophil count ≤1.0 x 109/L
   * ≥0.5 x 109/L and increasing following prior myelosuppressive treatment will be eligible
   * Screening Period 1 Only: Absolute lymphocyte count ≤1.0 x 109/L for solid tumor patients or ≤7.0 x 108/L for lymphoma patients prior to the apheresis procedure.
   * Platelet count ≤75 x 109/L absent platelet transfusion for 2 weeks
   * Hemoglobin (Hgb) ≤9 g/dL absent RBC transfusion for 2 weeks
   * ≥8 g/dL and increasing following prior myelosuppressive treatment will be eligible
   * Coagulation (prothrombin time [PT] or international normalized ratio [INR] and partial thromboplastin time [PTT] or activated partial thromboplastin time [aPTT])
   * >1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT/INR and PTT/aPTT is within therapeutic range of intended use of anticoagulants
   * Potassium, magnesium, calcium or phosphate abnormality > CTCAE v5.0 Grade 1 despite appropriate oral replacement therapy
   * Screening Period 1 Only: Serum triglycerides >500 mg/dL due to potential interference with cell separation methods
7. Impaired cardiac function or clinically significant cardiac disease, including any of the following:

   * Clinically significant and/or uncontrolled heart disease such as congestive heart failure requiring treatment (New York Heart Association [NYHA] Grade ≥2), uncontrolled hypertension, or clinically significant arrhythmia
   * Acute myocardial infarction or unstable angina pectoris <6 months prior to study entry
8. Patients with active, known or suspected autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs).

   1. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
   2. Patients with vitiligo, type 1 diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
9. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
10. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
11. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.

    Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
12. Has a known history of human immunodeficiency virus (HIV) infection. No HIV testing is required unless mandated by local health authority.
13. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.

    Note: No testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
14. Malignant disease, other than that being treated in this study expected to interfere with the assessment of efficacy in the opinion of the investigator.
15. Active infection requiring systemic therapy.
16. Patients requiring chronic treatment with systemic steroid therapy, other than replacement dose steroids in the setting of adrenal insufficiency. Topical, inhaled, nasal, or ophthalmic steroids are allowed.
17. Patients receiving systemic treatment with any immunosuppressive medication.
18. Use of any live vaccines against infectious diseases within 30 days of initiation of study treatment. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
19. Major surgery within 4 weeks of the first dose of study treatment (mediastinoscopy, insertion of a central venous access device, and insertion of a feeding tube are not considered major surgery).

    Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
20. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

    Note: Patients who have entered the follow-up phase of another investigational study may participate in this study as long as it has been 4 weeks after the last dose of the previous investigational agent.

    Note: Patients may participate in other local biomarker studies following documented discussion and approval from Repertoire Immune Medicines.

    Note: T-cell imaging agents may be permitted following documented discussion and approval with the Sponsor.
21. Presence of ≥CTCAE v5.0 Grade 2 toxicity from prior therapy (except alopecia, peripheral neuropathy, and ototoxicity, which are excluded if ≥CTCAE v5.0 Grade 3) due to prior cancer treatment.
22. Initiation of hematopoietic colony-stimulating growth factors (e.g. Granulocyte Colony Stimulating Factor [G-CSF], Granulocyte Macrophage Colony Stimulating Factor [GMCSF], Macrophage Colony Stimulating Factor [M-CSF]) ≤2 weeks prior to start of study drug. An erythroid stimulating agent is allowed as long as it was initiated at least 2 weeks prior to the first dose of study treatment.
23. An unresolved AE (must be ≤Grade 1 or the patient's baseline).
24. Prior treatment with CAR-T-cell therapy.
25. Has undergone prior allogeneic HSCT
26. RPTR-147 Monotherapy: Patients who were required to discontinue PD-1/PD-L1, CTLA-4, or other immunomodulatory antibodies due to ≥Grade 3 irAE may be included following discussion with the Sponsor.
27. RPTR-147:1 in Combination with pembrolizumab: Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137) and was discontinued from that treatment due to a Grade 3 or higher irAE.
28. Patients with a history of >3 lines of chemotherapy in the metastatic setting may be eligible for enrollment following discussion with the Sponsor.
29. Patients with a history of rapidly progressing disease on immunotherapy.

    1. Prior clinical or radiological disease progression (excluding pseudoprogression) within 8 weeks after starting prior immunotherapy with PD-1/PDL-1, CTLA-4 inhibitors.
    2. These patients may only be enrolled following discussion with the Sponsor to account for manufacturing time.
30. Prior therapy with PD-1/PDL-1, CTLA-4 or other immunomodulatory antibodies inhibitors:

    1. ≤2 weeks prior to the apheresis procedure
    2. ≤4 weeks prior to the first dose of study treatment
31. Systemic anti-cancer therapy within 5 half-lives or 2 weeks; whichever occurs first, of the apheresis procedure and the first dose of study treatment.

    1. Systemic cytotoxic agents that have major delayed toxicity, e.g. mitomycin C and nitrosoureas, ≤6 weeks prior to the first dose of study treatment
    2. Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible.
32. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
33. Has known psychiatric or substance abuse disorders that would interfere with cooperating with the requirements of the study.
34. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 150 days after the last dose of study treatment.
35. Women of childbearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during study treatment and for 120 days after the last dose of study treatment. Highly effective contraception methods include:

    1. Female sterilization, total hysterectomy, or tubal ligation at least 6 weeks before taking study treatment.
    2. Male sterilization (at least 6 months prior to screening). For female patients on the study the vasectomized male partner should be the sole partner for that patient.
    3. Use of oral (estrogen and progesterone), injected or implanted combined hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS) or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example, hormone vaginal ring or transdermal hormone contraception.

    In case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

    Women are considered post-menopausal and not of childbearing potential if they have had 12 months of natural amenorrhea with an appropriate clinical profile or have had surgical bilateral oophorectomy or tubal ligation at least 6 weeks prior to the first dose of study treatment.
36. A WOCBP who has a positive urine pregnancy test (e.g. within 72 hours) prior to treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects with dose limiting toxicities | At the end of cycle 1 (Each cycle is 28 days)
  Safety of RPTR-147:1 as a monotherapy
Number of subjects with dose limiting toxicities | At the end of cycle 1 (Each cycle is 21 days)
  Safety of RPTR-147:1 in combination with pembrolizumab
Number of subjects with dose limiting toxicities | At the end of cycle 1 (Each cycle is 21 days)
  Safety of RPTR-147:2 as a monotherapy
Frequency of dose interruptions | At the end of cycle 1 (Each cycle is 28 days)
  Tolerability of RPTR-147:1 as a monotherapy
Frequency of dose interruptions | At the end of cycle 1 (Each cycle is 21 days)
  Tolerability of RPTR-147:1 in combination with pembrolizumab
Frequency of dose interruptions | At the end of cycle 1 (Each cycle is 21 days)
  Tolerability of RPTR-147:2 in patients with HPV positive tumors

SECONDARY OUTCOMES:
Best overall response | Baseline through approximately 6 months after RPTR-147 last dose as monotherapy and in combination with pembrolizumab
  Per modified RECIST v1.1 (solid tumor) or Lugano classification (lymphoma)
Progression free survival | Baseline through approximately 6 months after RPTR-147 last dose as monotherapy and in combination with pembrolizumab
  Per modified RECIST v1.1 (solid tumor) or Lugano classification (lymphoma)
Maximum observed serum concentration of RPTR-147 as monotherapy and in combination with pembrolizumab | Baseline through approximately 1 year
  Maximum observed serum concentration
Area under the serum concentration-time curve | Baseline through approximately 1 year
  Area under the serum concentration-time curve
Immunogenicity of RPTR-147 as monotherapy and in combination with pembrolizumab | Pre-dose through approximately 1 year after RPTR-147/Pembrolizumab last dose
  Number of subject with anti-RPTR-147/Pembrolizumab antibodies

CONTACTS AND LOCATIONS:
Overall Officials: David Spriggs, MD, Study Director — Repertoire Immune Medicines
Locations (7):
- United States (7):
  - City of Hope, Duarte, California
  - Yale Cancer Center, New Haven, Connecticut
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No